CLINICAL TRIAL: NCT01232218
Title: Effectiveness of a Three-Dimensional Scapular-Humeral Mobilization Technique on Hemiplegic Shoulder Pain
Brief Title: Treatment Protocol for Hemiplegic Shoulder Pain
Acronym: TPHSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: University of Toronto (Other); Connect Learning Centre (Unknown); Ontario Stroke Network (Other)
Responsible Party: Principal Investigator, Denyse Richardson, Dr. Denyse Richardson, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRLP-10-010
Record Dates: First submitted 2010-10-25; First posted 2010-11-02 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Stroke; Hemiplegia; Shoulder Pain
Keywords: Cerebral Vascular Accident; Stroke; Hemiplegic; Shoulder pain; range of motion; scapula; mobilization
MeSH Terms: conditions — Stroke; Hemiplegia; Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current Standard Treatment (Active Comparator): Current standard treatment for hemiplegic shoulder pain will be provided to this group.
  Interventions: Other: Standard education/exercises for hemiplegic shoulder pain
- Standard treatment + study technique (Experimental): Participants will receive current standard treatment for hemiplegic shoulder pain PLUS an additional stretching/strengthening technique. Both groups will be allotted the same treatment time.
  Interventions: Other: Three dimensional Scapular-Humeral Mobilizations

INTERVENTIONS:
Other: Standard education/exercises for hemiplegic shoulder pain — Each participant will receive standard education for safe positioning and movement of the painful hemiplegic shoulder. Participants will also be provided with standard stretching and strengthening exercises by and experienced Occupational Therapist who will grade the level of exercise to suit their needs. Intervention will take place 3x/week for 1 hour.
  Other Names: Current Standard Treatment
  Arms: Current Standard Treatment
Other: Three dimensional Scapular-Humeral Mobilizations — Each participant will receive standard education for safe positioning and movement of the painful hemiplegic shoulder. Participants will also be provided with stretching and strengthening exercises by and experienced Occupational Therapist who will grade the level of exercise to suit their needs. Intervention will take place 3x/week for 1 hour. Participants in this group will receive an additional scapular humeral mobilization while simultaneously performing the standard stretching/strengthening exercise protocol.
  Other Names: Three-Demensional Scapular-Humeral Mobilization Technique; 3-D Scapular-Humeral Mobilizations
  Arms: Standard treatment + study technique

SUMMARY:
The purpose of this study is to determine if a specific stretching and strengthening protocol, in addition to current standard treatment, is more effective for treating post-stroke shoulder pain than current standard treatment alone.

DETAILED DESCRIPTION:
Current standard treatment of post-stroke shoulder pain includes joint protection (i.e., slings and protective positioning) and stretching/strengthening exercises through a pain-free range. Although the added movement of the shoulder blade when moving the post-stroke arm has been recommended in the literature, no studies to date have been found which directly looks at the impact of providing synchronized three-dimensional scapular and humeral movement during therapy. Due to the integral relationship between the scapula and the humerus during movement, it is hypothesized that an increase in 3-dimensional shoulder blade mobility in the painful post-stroke shoulder will contribute to increased pain-free 3-dimensional arm movement. This double-blind randomized-controlled study aims to investigate the effectiveness of this 3-D approach at addressing post-stroke shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of shoulder pain secondary to altered alignment and/or neuro-muscular movement patterns post-stroke;
* medically stable and 2-24 months post onset of stroke;
* between stages of 2-5 of the Chedoke-McMaster stages of upper extremity motor recovery;
* not currently receiving any other active neuro-rehabilitation intervention to promote stroke recovery;
* cognitively able to provide informed consent, follow specific testing commands, and communicate their level of pain during assessment and treatment.

Exclusion Criteria:

* a history of shoulder pain prior to the onset of the stroke;
* shoulder pain which is secondary to any history of trauma, fractures, arthritis or joint instability of the neck, spine, ribs, or shoulder girdle before or after the stroke; possible rotator cuff tears;
* shoulder-hand syndrome; thalamic or central pain; spinal cord pathology; osteoporosis;
* any medical condition which may affect the ability to participate in an active rehabilitation exercise program (i.e., uncontrolled hypertension or angina).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Measurement of active and passive pain-free shoulder range of motion | 1 week prior to intervention
  Using a 3-dimensional motion capture system and digitizer system, we will determine degrees of pain-free active and passive movement of the shoulder and arm for each participant. Changes in range of motion between pre and post-treatment will be calculated.
Measurement of active and passive pain-free shoulder range of motion | 1 week after intervention
  Using a 3-dimensional motion capture system and digitizer system, we will determine degrees of pain-free active and passive movement of the shoulder and arm for each participant. Changes in range of motion between pre and post-treatment will be calculated.
Measurement of active and passive pain-free shoulder range of motion | one month after intervention
  Using a 3-dimensional motion capture system and digitizer system, we will determine degrees of pain-free active and passive movement of the shoulder and arm for each participant. Changes in range of motion between pre and post-treatment will be calculated.

SECONDARY OUTCOMES:
Visual Analogue Scale (used to report the degree of pain experienced during different levels of functional reaching) | 1 week prior to intervention
  Participants will be asked to subjectively rate their level of pain (on a scale of 1-10) when progressively reaching to the top of the head and behind the back.
Chedoke McMaster Pain Inventory | 1 week prior to intervention
  A descriptive scale for quantifying hemiplegic shoulder pain
Visual Analogue Scale (used to report the degree of pain experienced during different levels of functional reaching) | 1 week after intervention
  Participants will be asked to subjectively rate their level of pain (on a scale of 1-10) when progressively reaching to the top of the head and behind the back.
Chedoke McMaster Pain Inventory | 1 week after intervention
  A descriptive scale for quantifying hemiplegic shoulder pain
Visual Analogue Scale (used to report the degree of pain experienced during different levels of functional reaching) | 1 month after intervention
  Participants will be asked to subjectively rate their level of pain (on a scale of 1-10) when progressively reaching to the top of the head and behind the back.
Chedoke McMaster Pain Inventory | 1 month after intervention
  A descriptive scale for quantifying hemiplegic shoulder pain

CONTACTS AND LOCATIONS:
Overall Officials: Denyse Richardson, MD; M.Ed, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada